CLINICAL TRIAL: NCT06462495
Title: Head-to-head Comparison of [18F]F-PSMA-N5 With [18F]F-PSMA-1007 PET/CT in Prostate Cancer Diagnosis, Recurrence, and Metastasis: a Prospective Study
Brief Title: Head-to-head Comparison of [18F]F-PSMA-N5 With [18F]F-PSMA-1007 PET/CT in PCa Diagnosis, Recurrence, and Metastasis
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PSMA PET STUDY -01
Record Dates: First submitted 2024-06-12; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Prostate Cancer; PET/CT
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [18F]F-PSMA-N5 and [18F]F-PSMA-1007 PET/ CT scan (Experimental): Subjects PET/CT imaging: On any two days for two consecutive weeks, each subject underwent a PET/ CT scan after intravenous injection of [18F]F-PSMA-N5 and [18F]F-PSMA-1007.
  Interventions: Drug: [18F]F-PSMA-N5; Drug: [18F]F-PSMA-1007

INTERVENTIONS:
Drug: [18F]F-PSMA-N5 — Each subject receive a single intravenous injection of [18F]F-PSMA-N5, and undergo PET/CT imaging within the specificed time.
  Other Names: [18F]F-PSMA-N5 injection
Drug: [18F]F-PSMA-1007 — Each subject receive a single intravenous injection of [18F]F-PSMA-1007, and undergo PET/CT imaging within the specificed time.
  Other Names: [18F]F-PSMA-1007 injection

SUMMARY:
To prospectively evaluate the radiodrug biodistribution of a novel PET imaging agent [18F]F-PSMA-N5 in different organs of prostate cancer patients and its diagnostic efficacy in the diagnosis, recurrence and metastasis of prostate cancer, and to compare with [18F]F-PSMA-1007.

DETAILED DESCRIPTION:
[18F]F-PSMA-N5 PET/CT was used for initial assessment of prostate cancer or detection of recurrence. The maximum standardized uptake value (SUVmax) was used to evaluate tumor uptake. The sensitivity, specificity, the number and accuracy of lesions identified and the distribution of lesions in each organ were calculated and compared with those of [18F]F-PSMA-1007 PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* Aged from 18 to 90 years old;
* Complete MRI images and clinical data (such as PSA level, Gleason grade, etc.);
* Prostate cancer detected by PSA or imaging examination, or clinically suspected recurrence after standardized treatment;
* simultaneous [18F]F-PSMA-N5 and [18F]F-PSMA-1007 examinations within two weeks;
* Willing to undergo surgery or needle biopsy for pathological examination after examination, or confirmed as prostate cancer by histopathology before or after treatment;
* Sign informed consent.

Exclusion Criteria:

* Patients who cannot cooperate with the examination;
* Concurrent malignant tumors;
* Previous alcohol allergy;
* Patients with liver and kidney dysfunction;
* Other circumstances deemed by the investigator to be inappropriate for trial participation.

Ages: 18 Years to 90 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Standard uptake value(SUV) | 30 days
  Standard uptake value(SUV) of [18F]F-PSMA-N5 and [18F]F-PSMA-1007 for each target lesion of subjects.

SECONDARY OUTCOMES:
Diagnostic efficacy | 30 days
  The sensitivity, specificity and accuracy of [18F]F-PSMA-N5 and [18F]F-PSMA-1007 PET/CT were calculated.
Number of lesions | 30 days
  The number of lesions detected by [18F]F-PSMA-N5 and [18F]F-PSMA-1007 PET/CT.

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Xie, Study Chair — The First Affiliated Hospital of USTC (Anhui Provincial Hospital)
Locations (1):
- The First Affiliated Hospital of China University of Science and Technology（Anhui Provincial Hospital）, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No